CLINICAL TRIAL: NCT01374139
Title: A Phase 1, Open-Label, Randomized, Single-Dose, 2-Cohort, 2-Way Crossover Bioequivalence Study To Compare The Bosutinib Clinical Tablet And Clinical Capsule And To Investigate Food Effect On Bosutinib Commercial Formulation in Healthy Subjects
Brief Title: Bioequivalence And Food Effect Study Of Bosutinib In Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B1871035
Record Dates: First submitted 2011-06-07; First posted 2011-06-15 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Philadelphia Chromosome Positive (Ph+) Chronic Myeloid Leukemia (CML)
Keywords: Bosutinib; Bioequivalence and Food Effect Studies
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: Bosutinib
- Cohort 2 (Experimental)
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib — 5 clinical 100 mg tablets and 100 mg capsules, 500 mg, single dose, 2x2 crossover under fed condition
  Other Names: SKI-606, PF-05208763
  Arms: Cohort 1
Drug: Bosutinib — 4 commercial 100 mg tablets, 400 mg, single dose, 2x2 crossover under fed/fast condition
  Other Names: SKI-606, PF-05208763
  Arms: Cohort 2

SUMMARY:
The purpose of this study is to demonstrate the bioequivalence of the clinical tablet formulation (100 mg x 5) to the clinical capsule formulation (100 mg x 5) in healthy subjects under fed condition (Cohort 1) and to investigate the effect of a high-fat meal on the pharmacokinetics of bosutinib after administration of the proposed commercial tablet formulation (100 mg x 4) in healthy subjects (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female of non childbearing potential subjects between the ages of 21 and 55 years, inclusive.
* Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12 Lead ECG or clinical laboratory tests.

Exclusion Criteria:

* Pregnant or nursing women or women of childbearing potential.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Plasma Cmax for bosutinib. | 96 hr post dose in each period
AUCt for bosutinib. | 96 hr post dose in each period
Plasma AUCinf for bosutinib. | 96 hr post dose in each period
AUClast for bosutinib. | 96 hr post dose in each period
Tmax for bosutinib. | 96 hr post dose in each period
t½ for bosutinib. | 96 hr post dose in each period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1871035&StudyName=Bioequivalence%20And%20Food%20Effect%20Study%20Of%20Bosutinib%20In%20Healthy%20Subjects